CLINICAL TRIAL: NCT04774887
Title: ERADICATING CERVICAL CANCER IN KENYA: Benefits of Community-based Prevention, and the Effects of Aflatoxin on HPV Vaccination (MISP 60403) (MISP2)
Brief Title: ERADICATING CERVICAL CANCER IN KENYA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Moi University (Other)
Responsible Party: Principal Investigator, Darron Brown MD, MPH, Professor of Medicine, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 60403
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Human Papilloma Virus; HIV Infections
Keywords: HPV; HIV; Kenya
MeSH Terms: conditions — HIV Infections | interventions — Papillomavirus Vaccines

STUDY DESIGN:
Intervention Model Description: Children of mothers in the study will receive the HPV vaccine as per Kenya guidelines.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HPV vaccination (Experimental): Children receiving HPV vaccine will be studies for seroconversion to HPV types, and aflatoxin levels in blood will be measured and compared to seroconversion.
  Interventions: Biological: HPV vaccine, Merck

INTERVENTIONS:
Biological: HPV vaccine, Merck — Vaccination against HPV will be offered to 900 children/grandchildren aged 9 through 18 of women attending the Community Meetings.

SUMMARY:
This is a study of a strategy designed to 1) increase cervical cancer screening using a community-based approach, and 2) determine the efficacy of HPV vaccination in a region of Kenya where half of all children are chronically exposed to aflatoxin.

DETAILED DESCRIPTION:
Cervical cancer is caused by oncogenic HPV, and is the main cause of cancer-related death among Kenyan women. This malignancy is preventable through a combination of screening of adult women and vaccination of children and adolescents against HPV infection. However, only 5% of Kenyan women are regularly screened, and only 14% have ever been screened, which in Kenya is done by a method known as Visual Inspection with Acetic Acid (VIA). Obstacles to screening include travel to clinics, costs, poor specificity of VIA, lack of trained personnel, and others. In addition, while safe and effective HPV vaccines have been available for 15 years, very few (<1%) Kenyan children and adolescents have been vaccinated. Obstacles to vaccination include costs, delivery infrastructure, lack of education, travel to clinics, and others. In addition, there are few studies of HPV vaccination in African children, and two-dose regimens may not provide adequate protective antibody levels among children chronically exposed to aflatoxin, a potent immunosuppressive agent found in contaminated corn. Investigators propose a study of a strategy designed to 1) increase cervical cancer screening using a community-based approach, and 2) determine the efficacy of HPV vaccination in a region of Kenya where half of all children are chronically exposed to aflatoxin.

Objective 1 (Cervical cancer screening): Evaluate High-Risk (HR)-HPV DNA testing of self-collected vaginal swabs as a triage step for VIA among rural Kenyan women.

Hypothesis: All women with negative HR-HPV DNA tests will have normal VIA examinations or falsely-abnormal VIA examinations based on cervical biopsy results. The rationale is that if this hypothesis is correctly proven, it will suggest that VIA is unnecessary for women with negative HR-HPV DNA tests in self-collected vaginal swabs.

Objective 2 (HPV vaccination): Determine the effects of chronic aflatoxin exposure among Kenyan children/adolescents on the likelihood of seroconversion to HPV types represented in the HPV vaccine.

Hypothesis: Compared to children/adolescents without detectable plasma aflatoxin, children/adolescents with evidence of chronic aflatoxin exposure will have a reduced likelihood of seroconversion to HPV types represented in the HPV vaccine. The rationale is that if this hypothesis is correctly proven, it will suggest that adjustments in vaccination doses/schedules may be needed for children with chronic exposure to aflatoxin to assure adequate protection against HPV infection.

ELIGIBILITY:
Inclusion Criteria:

* Kenyan women between ages of 18 and 60 years and children/grandchildren aged 9 through 18 of women attending the Community Meetings.

Exclusion Criteria: Pregnancy, history of cervical cancer, allergy to HPV vaccine (children)

-

Ages: 9 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2021-11-13 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
Detection of high-grade cervical intraepithelial neoplasia (CIN) 2/3+ | Two years
  Rate and relative risk of biopsy-proven VIA abnormality between women with positive HR-HPV and women with negative HR-HPV.
Seroconversion to all HPV vaccine types | Two years
  Rate and relative risk of seroconversion to all HPV types combined and to each of the nine HPV types represented in the nine-valent HPV vaccine between children with and without plasma aflatoxin detection.

CONTACTS AND LOCATIONS:
Locations (1):
- Webuye Clinic, Webuye, Kenya

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data will be available on request to researchers.